CLINICAL TRIAL: NCT07150117
Title: Evaluating the Acceptability of a Cycling-Based Aerobic Exercise Intervention for Individuals With Chemotherapy-Induced Peripheral Neuropathy (CIPN): A Proof-of-Concept Study
Brief Title: Cycling-Based Aerobic Exercise Intervention for Individuals With Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Acronym: CYCLE-CIPN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-25-0188
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Adults
Keywords: peripheral neuropathy; chemotherapy; exercise; aerobic; cancer
MeSH Terms: conditions — Neoplasms; Peripheral Nervous System Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Proof of concept study
Masking Description: An independent assessor will be used to collect post-intervention outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerobic exercise intervention (Experimental): Cycling-based aerobic exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — A supervised 12-week cycling-based aerobic exercise intervention performed twice per week.

SUMMARY:
CYCLE-CIPN is a proof-of-concept study designed to evaluate whether a prescribed aerobic exercise intervention has the potential to reduce the symptoms and functional impact of CIPN. The small number of participants in the proposed study will allow us to make decisions on the feasibility ("go/no-go") of a future larger-scale trial.

The protocol will assess feasibility and acceptability through recruitment, completion, adherence, program satisfaction, and safety. The study will also evaluate CIPN symptoms using both patient-reported and objective outcome measures, as well as fitness and quality of life outcomes. We aim to recruit 30 participants.

The Health Research Board of Alberta Cancer Committee has approved this study. Participants will participate in a stationary cycling-based aerobic exercise program biweekly for 12 weeks. Exercise sessions will be supervised and progressive, between 30 and 60 minutes each.

DETAILED DESCRIPTION:
CIPN is a common and dose-limiting side effect of neurotoxic chemotherapeutic agents used in cancer treatments, with symptoms affecting up to 100% of patients depending on the drug class. These symptoms-classified as positive (e.g., tingling, pain, allodynia) or negative (e.g., numbness, decrease in fine motor skills) -primarily occur in the hands and feet. CIPN persists in approximately 30% of patients six months post-treatment, significantly impacting quality of life. As there are no pharmacological treatments established for CIPN, there is a critical need to explore lifestyle interventions to improve survivorship care.

Exercise is a promising lifestyle intervention for managing CIPN, with research suggesting improvements in CIPN symptoms such as pain and numbness. Most existing studies have utilized multimodal exercise interventions (typically aerobic, resistance, and balance training) and often rely exclusively on patient-reported outcome measures (PROMs), limiting generalizability. There is significant variability in CIPN outcome measures used across studies, as a standardized core outcome set has not yet been established. Aerobic exercise may reduce CIPN symptoms through neurotrophins that affect neurons, peripheral nerves, and inflammation; however, the exact mechanisms remain unclear. While aerobic exercise shows considerable potential for CIPN symptom reduction, its isolated effects on CIPN-associated symptoms and function observed through the use of both PROMs and objective clinical measures remain unexplored. The FITT principle (Frequency, Intensity, Time, Type) provides a standardized framework for exercise prescription, yet few studies have examined its application in dosing CIPN-specific aerobic exercise interventions. Stationary cycling offers a safe, non-weight-bearing aerobic exercise mode that is accessible for individuals with CIPN. To address current research gaps, further investigation is warranted to examine the feasibility, acceptability, and outcomes of cycling-based aerobic exercise intervention using both patient-reported and objective outcome measures.

The primary objective of this study is to determine the feasibility and acceptability of a stationary cycling-based aerobic exercise program for individuals with CIPN using both objective and patient-reported outcome measures, as defined by:

Recruitment rate: 30 participants recruited within one year

Completion rate: >70% of participants consenting to the study complete the 12-week assessment

Adherence rate: average completion of >70% of the FITT prescription variables

Program satisfaction: >70% reporting high to very high program satisfaction

Safety: no serious adverse events related to exercise

The study will involve 30 participants (aged 18+) with CIPN, either undergoing or post-chemotherapy. Participants will be recruited from the Cross Cancer Institute and the University of Alberta's Cancer Rehabilitation Clinic. Subjects will be screened for eligibility, and if all eligibility criteria are met, they will be provided with a study brochure. Participants will be asked to contact the investigators if they are interested. All participants are required to provide written informed consent as per the Health Research Ethics Board of Alberta: Cancer Committee (HREBA-CC).

The intervention consists of a 12-week aerobic exercise stationary cycling program to determine the acceptability and appropriateness of the intervention for CIPN. The program will be administered through the Cancer Rehabilitation Clinic and Exercise Oncology Research Laboratory at the University of Alberta. Based on the results of the participants' baseline assessments (i.e. % heart rate maximum from cardiopulmonary exercise testing), participants will receive individualized exercise programs. Twice weekly, participants will attend in-person small group exercise sessions, supervised by certified exercise physiologists and qualified exercise professionals (supervisor-to-participant ratio of 1:3). Exercise prescriptions were adapted from the most recent exercise guidelines for cancer survivors and previous aerobic-exercise-including trials in individuals with cancer. Each week, participants will undergo two different exercise sessions: (1) continuous cycling-based aerobic exercise, and (2) high-intensity interval training (HIIT) on a cycle ergometer.

Analyses: All participants who provide informed consent and complete the baseline assessment will be considered for analysis. A per-protocol (PP) analysis will be implemented as there is no randomization or multi-group designation in this study. Participants included in the PP analysis will be those who provide informed consent, complete both pre- and post-intervention assessments, and attend at least 70% of exercise sessions. Participants who do not meet the PP analysis criteria will be excluded from the PP analysis, but will be included in proof-of-concept outcomes (i.e. completion rate, adherence, adverse events). Descriptive statistics will be used to summarize demographic characteristics. Completion, recruitment, and adherence rates will be calculated using numbers and percentages, and the mean rates will be reported. All statistical analyses in the PP analysis will use a two-tailed, repeated measures t-test with a significance level set at α=0.05. Effect size (i.e. Cohen's d) will be reported to describe the magnitude of change between pre- and post-intervention assessments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Cancer diagnosis stage I to III
* CIPN: grade 1 (mild)
* Receiving or have received chemotherapy treatment for cancer
* Speak, read and understand English

Exclusion Criteria:

* Medical conditions that cause additional neuropathy symptoms (i.e. diabetes)
* Any uncontrolled medical conditions
* Will undergo surgery or radiation therapy during the study period
* Are already receiving an aerobic exercise training program
* Are already participating in an exercise-based research study
* Are unable to provide signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment | One year
  Recruitment rate of 30 participants in one year

SECONDARY OUTCOMES:
Study completion | One year
  Completion rate: >70% of participants consenting to the study complete the 12-week assessment
Adherence | 12 weeks
  Adherence rate >70% for the prescription variables
Program satisfaction | 12 weeks
  >70% of participants reporting high to very high program satisfaction with higher scores indicating higher satisfaction with the intervention, program delivery and perceived benefits.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L McNeely, PhD, Principal Investigator — University of Alberta

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available no later than 12 months following primary publication of study findings.
  Data will be deposited and made accessible through Borealis, the Canadian Dataverse Repository (https://borealisdata.ca), a secure platform for sharing research data. Access will be granted via request through the repository, subject to approval and under a data sharing agreement outlining the terms of use and protection of participant privacy.
Supporting Information: CSR
Time Frame: Data will be made available no later than 12 months following primary publication of study findings.
Access Criteria: Data will be shared on request with qualified researchers affiliated with academic institutions, healthcare organizations, or other not-for-profit entities conducting methodologically sound research.
URL: https://borealisdata.ca